CLINICAL TRIAL: NCT05062356
Title: Prospective Randomized Study Comparing Suprainguinal Fascia Iliaca Block vs. Pericapsular Nerve Group Block vs. Local Anesthetic Infiltration vs. Spinal Anesthetic Without Adjuncts for Pain Control Following Total Hip Arthroplasty
Brief Title: Pain Control Following Total Hip Arthroplasty
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Mary's Research Center, Canada (Other)
Responsible Party: Principal Investigator, Anthony Albers, MD, MD, Orthopaedic Surgeon, St. Mary's Research Center, Canada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMHC - 21- 02
Record Dates: First submitted 2021-09-20; First posted 2021-09-30 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Chronic Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Epinephrine; Prilocaine; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Suprainguinal fascia iliaca compartment block (FICB) (Experimental): Suprainguinal fascia iliaca compartment block (FICB) is a technique that involves injection of local anesthetics underneath the fascia of the iliacus muscle to block the femoral nerve, the lateral femoral cutaneous nerve and, possibly, the obturator nerve.
  Interventions: Drug: Bupivacaine Hydrochloride 0.25% Injection Solution_#2; Drug: EPINEPHrine 1:200,000 / Prilocaine HCl 4 % 1.8 ML Cartridge; Drug: Ketorolac
- Pericapsular nerve group block (PENG) (Active Comparator): The pericapsular nerve group block (PENG) is a technique that involves injection of local anesthetic in the musculofascial plane between the psoas muscle and the superior pubic ramus.
  Interventions: Drug: EPINEPHrine 1:200,000 / Prilocaine HCl 4 % 1.8 ML Cartridge; Drug: Bupivacaine Hydrochloride 0.5% Injection Solution_#2; Drug: Ketorolac
- Local analgesia infiltration (LAI) (Sham Comparator): local anesthetic infiltration (LAI) into the anterior pericapsular tissues
  Interventions: Drug: Bupivacaine Hydrochloride 0.25% Injection Solution_#2; Drug: EPINEPHrine 1:200,000 / Prilocaine HCl 4 % 1.8 ML Cartridge; Drug: Ketorolac
- No adjunct: spinal anaesthesia (control) (Sham Comparator): Standard spinal anesthesia technique
  Interventions: Drug: Bupivacaine Hydrochloride 0.5% Injection Solution_#2; Drug: Ketorolac

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride 0.25% Injection Solution_#2 — 40cc
  Arms: Local analgesia infiltration (LAI); Suprainguinal fascia iliaca compartment block (FICB)
Drug: EPINEPHrine 1:200,000 / Prilocaine HCl 4 % 1.8 ML Cartridge — 10cc
  Arms: Local analgesia infiltration (LAI); Pericapsular nerve group block (PENG); Suprainguinal fascia iliaca compartment block (FICB)
Drug: Bupivacaine Hydrochloride 0.5% Injection Solution_#2 — 20cc
  Arms: No adjunct: spinal anaesthesia (control); Pericapsular nerve group block (PENG)
Drug: Ketorolac — 15mg

SUMMARY:
Total hip arthroplasty (THA) is one of the most common surgical procedures performed in elderly patients, with its main indication being end-stage osteoarthritis of the hip1. It is estimated that over 572,000 patients per year will undergo THA in the USA alone by 20301 and postsurgical pain associated with THA remains a significant issue. Postoperative pain is associated with delayed joint mobilization, ambulation, patient satisfaction and can often delay the patient's discharge home1.

Multimodal analgesia for the management of postoperative pain following THA is now standard of care2,3. It involves a combination of local anesthetic infiltration (LAI), peripheral nerve blocks (PNBs), analgesics such as non-steroidal anti-inflammatory drugs (NSAIDs), acetaminophen and/or other medications, including gabapentinoids and opioids. Using multiple analgesic modalities allows for an easier and faster recovery for THA patients and ultimately allows for reduction in postoperative narcotic use and it's associated negative side effects. Total hip arthroplasty can be performed under either general anesthesia, epidural anesthesia or most commonly under spinal anesthesia, with or without epidural morphine. The adjunctive use of LAI, pericapsular nerve group (PENG) block or suprainguinal fascia iliaca compartment block (FICB) for postoperative pain management is becoming more widespread, although evidence on their efficacy has been inconsistent4-8. As such, comparative evaluation of these adjuctive analgesic modalities is imperative to optimize postoperative pain management following THA.

DETAILED DESCRIPTION:
Suprainguinal fascia iliaca compartment block (FICB) is a technique that involves injection of local anesthetics underneath the fascia of the iliacus muscle to block the femoral nerve, the lateral femoral cutaneous nerve and, possibly, the obturator nerve9. The pericapsular nerve group block (PENG) is a technique that involves injection of local anesthetic in the musculofascial plane between the psoas muscle and the superior pubic ramus. Evidence to date shows that FICB and PENG may be effective modalities to provide postoperative pain control following THA and could reduce opioid consumption10. The above procedures have been documented as safe and effective when performed by a qualified anesthetist but come with various risks (potential motor / sensory blocade especially) and associated cost. Alternatively, or in conjunction to the above procedures, the orthopedic surgeon can perform local anaesthetic infiltration (LAI) into the anterior pericapsular tissues. To date, no study has compared the efficacy of FICB, PENG block and LAI in a randomized study, therefore a preferred postoperative analgesic regimen has yet to be determined.

In this randomized trial, the investigators aim to evaluate postoperative pain and side effects related to pain control in patients who receive FICB versus LAI versus PENG block following THA. The investigators aim to compare these procedures between each other and assertain whether these techniques compare favourably to spinal anesthetic as a control group.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old) who require an inpatient primary total hip arthroplasty under spinal anesthesia
* Written consent
* Any gender

Exclusion Criteria:

* Patients who require revision surgery
* Anesthesia other than spinal (general, epidural, other)
* Body mass index (BMI) > 45 kg/m2
* Allergies to study medication
* Previous fracture to affected area
* Previous surgery to the affected hip
* Diagnosis other than osteoarthritis (avascular necrosis, significant deformity such as post-Perthes, slipped capital femoral epiphysis, dysplasia classified as Crowe 3 or 4, or other diagnoses causing significant deformity of the femoral head or acetabulum)
* THA for hip fractures
* Patients taking daily opiod analgesics pre-operatively
* Anesthetist on day of surgery who does not perform FICB and PENG and no alternate anesthetist available to perform the block
* Patients who do not understand, read or communicate in either French or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Visual analog pain scale (VAS) | At 4 hours
  The primary outcome was chosen as VAS at 4 hours post-op. The investigators debated between VAS score and narcotic consumption, as both have their limitations. VAS score, which is used as primary outcome in most similar studies1, 4-9 can be affected by narcotic consumption and vice-versa. Narcotic consumption is also variable given the need for patients to ask for the medication (with the subjective nature of pain tolerance) and requirement that nursing be available to administer it while in hospital. Some studies have attempted to circumvent these limitations by utilizing patient controlled analgesia (PCA) pumps. The researchers wanted to avoid this because it does not reflect current clinical practice. Therefore, VAS was chosen at 4 hours, a time frame where the spinal effect is likely diminished, the blocks are most effective, the need for breakthrough narcotics is low, being in line with the current literature

SECONDARY OUTCOMES:
Patient satisfaction with pain control | at 4 hours
  Secondary outcome measures include patient satisfaction with pain control at the above mentioned time points using a four point Likert scale, the need for breakthough opioids in the first 4 hours, the number of morphine equivalents consumed for the first 48 hours post-op and length of hospital stay. Complications related to anesthesia such as motor nerve block (femoral or sciatic), any perceived peripheral sensory changes, urinary retention, post-operative nausea/vomiting or signs/symptoms of local anaesthetic toxicity will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Anthony Albers, MDCM, FRCSC, Principal Investigator — McGill University, Department of Surgery
Locations (1):
- St. Mary's Hospital Center, Montreal, Quebec, Canada